CLINICAL TRIAL: NCT05908825
Title: A Split-Face, Double-Blind, Placebo-Controlled Study Assessing the Use of a Novel Exfoliative Serum With A Chemical Peel to Improve Photodamage
Brief Title: Placebo-Controlled Study Assessing the Use of a Novel Exfoliative Serum With A Chemical Peel to Improve Photodamage in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Institute for Clinical Research (Network)
Collaborators: SkinCeuticals (Unknown)
Responsible Party: Principal Investigator, Edward Lain, MD, Principal Investigator, Austin Institute for Clinical Research
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CATALYST-001
Record Dates: First submitted 2023-05-10; First posted 2023-06-18 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Photodamaged Skin
MeSH Terms: interventions — Ascorbic Acid; acetohydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 day application of study product A and B (Other): Subjects will be given study drug and instructed to topically apply to the treatment area, Study Product A or Study Product B, placebo serum or novel exfoliative serum, to the respectively randomized half of the face, once daily for 20 consecutive days.
  Interventions: Drug: Vitamin C with AHA Exfoliative Serum; Drug: Placebo serum
- 42 day application of study product A and B (Other): Subjects who the investigator decides to continue treatment at Day 21, will be given study drug and instructed to topically apply to the treatment area, Study Product A or Study Product B, placebo serum or novel exfoliative serum, to the respectively randomized half of the face, once daily for an additional 21 consecutive days.
  Interventions: Drug: Vitamin C with AHA Exfoliative Serum; Drug: Placebo serum

INTERVENTIONS:
Drug: Vitamin C with AHA Exfoliative Serum — Catalyst is a novel skincare product comprised of low concentrations of multiple hydroxy acids and will be randomly assigned as Product A or Product B to be applied to one side of the face.
  Other Names: Skinceuticals C + AHA
Drug: Placebo serum — Placebo serum will be randomly assigned as Product A or Product B to be applied to one side of the face.

SUMMARY:
This is a split-face, double-blind, placebo-controlled study assessing the use of a novel exfoliative serum with a chemical peel to improve photodamage in healthy female subjects between the ages of 30 and 65 years, inclusive, with Fitzpatrick skin types I-VI.

DETAILED DESCRIPTION:
A single-center study. Clinical efficacy will be assessed using the modified Griffith's scale. Instrumentation will be assessed using VISIA imaging procedures, and TEWL (transepidermal water loss). Tolerability will be assessed in subjects through objective tolerance grading and subjective tolerance assessment. In addition, subject perception of the product will be evaluated by questionnaires. Live investigator clinical efficacy grading, tolerance evaluations, and subject self-assessments; will be performed at baseline and Days 7, 14, 21, 31, and 42. Additionally instrumentation measurements of erythema and hyperpigmentation will be calculated by digital assessments of facial photographs.

All data will be collected by the clinical site and delivered to SGS in Excel files, including demographic information, clinical grading of efficacy and tolerability evaluations, Tewameter, and self-assessment questionnaire data. Data review and analyses will be performed by an independent data committee. Interim topline data will be sent to the Sponsor after Day 42. End-of-study topline data will be sent at 10 business days after study completion. A clinical study report will be drafted using an SGS report template and incorporating any documented Sponsor preferences on file with SGS. The draft report will be submitted to the Sponsor for approval prior to finalization, and revisions may be made at the Sponsor's request. SGS will submit the draft report to the Sponsor 20-30 business days after approval of all statistical analysis and receipt of study documents from the study site. Any additions and changes to the statistical analysis after study completion may delay issuance of the draft report. After receiving the draft report, the Sponsor will have 6 months to make revisions. If SGS has received no revisions or comments within 6 months, the report will be approved for finalization. Every effort will be made to send the final report to the Sponsor within 10 business days after Sponsor approval or after the 6-month period has passed.

A total of 25 subjects are planned to be enrolled. Subjects who met the specified inclusion/exclusion criteria will be randomized to receive the novel exfoliative serum on one side and placebo on the other side on Day 0 of the study. On Day 14 of the study, each subject will receive a chemical peel as deemed appropriate by the Investigator and based on Fitzpatrick skin type. The chemical peel will be either TCA SmartPeel or Micropeel 30, per Investigator prerogative based on subject's skin sensitivity. For subject with Fitzpatrick Skin Type of IV-VI will receive the Micropeel. Following the chemical peel all subjects will discontinue use of the placebo and novel exfoliative serum. On Day 21, facial skin will be examined by the Investigator in-office to determine if each subject may resume the Day 0 randomized treatment regimen. All evaluations will be done in a double-blind fashion. Clinical efficacy endpoints will be evaluated on Days 7, 14, 21, 31 and 42. Tolerance endpoints will be evaluated on Days 14, 21, 31 and 42. In addition, tolerability will be evaluated on Day 16 via tele-visit (phone call). Physician assessments, patient-reported outcomes, and digital assessments of photographs will be captured during this study.

A subject may be discontinued from study treatment at any time if the subject, the Investigator, or the Sponsor feels that it is not in the subject's best interest to continue. If a subject is withdrawn from treatment due to an AE, the subject will be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized.

All subjects who discontinue study treatment should come in for an early discontinuation visit as soon as possible and then should be encouraged to complete all remaining scheduled visits and procedures. All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. If a subject withdraws prior to or during the procedure, an additional subject may be enrolled to replace the withdrawn subject. The sponsor may elect to close the trial at any time during the course of the study. Any data collected prior to termination may be analyzed as specified in the protocol.

The Investigator will probe, via discussion with the subject, for the occurrence of AEs (adverse events) during each subject visit and record the information in the site's source documents. Adverse events will be recorded in the subject CRF (case report form). Adverse events will be described by duration (start and stop dates and times), severity, outcome, treatment and relation to study drug, or if unrelated, the cause. Study site will document all SAEs (serious adverse events) that occur (whether or not related to study treatment). The collection period for all SAEs will begin after informed consent is obtained and end after procedures for the final study visit have been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects aged between 30 and 65 years, inclusive
2. Fitzpatrick skin type I-VI
3. All skin types, including sensitive skin
4. Mild to moderate severity (score of 3 to 6; modified Griffiths scale) of the following attributes on the global face:

   1. Smoothness, tactile and visual
   2. Dark spot intensity
   3. Hyperpigmentation
   4. Clarity
   5. Radiance
   6. Skin tone evenness
   7. Firmness (visual)
   8. Elasticity (tactile)
   9. Overall healthy skin appearance
   10. Global fine lines
   11. Appearance of pores
5. No known medical conditions that, in the Investigator's opinion may interfere with study participation
6. Willingness to cooperate and participate by following study requirements
7. Individuals must sign an informed consent and a photography consent

Exclusion Criteria:

1. Subjects that are being treated for cancer or have a history of facial skin cancer on the test areas
2. Subjects with sunburn, moderate to pronounced suntan, pronounced asymmetric skin aging, tattoos, scars or other disfiguration, dilated vessels or other conditions on the test area that might influence the test results
3. Subjects currently taking certain medications which in the opinion of the Investigators may interfere with the study. This includes but not limited to routine high dosage use of anti-inflammatory drugs (aspirin, ibuprofen, corticosteroids [steroid nose drops, inhalers and/or eye drops are permitted]), and immunosuppressive drugs
4. Subjects with self-reported, uncontrolled systemic disease which, in the opinion of the Investigator, may hinder either the subject's ability to perform all responsibilities of the trial or the Investigator's ability to perform assessments
5. Women known to be pregnant, nursing or planning to become pregnant
6. Subjects participating in other facial clinical studies
7. Subjects who have routinely used an alpha-hydroxy-acid (AHA) or a beta-hydroxy-acid (BHA) containing product within two weeks or Retin-A, Retin-A Micro, Renova, Differin, Avita, Tazorac, or Soriatane within 8 weeks of the study start or have taken Isotretinoin within one year of the study start. Subjects who have used Retinol in the last 4 weeks
8. Subjects with current flaring moderate to severe inflammatory acne
9. Subjects who have had ablative laser treatments, microneedling, and/or chemical peels or dermabrasion within the last six months
10. Subjects who have had botulinum type-A toxin (e.g. Botox®, Dysport® or Xeomin ®) within the last 3 months
11. Subjects who have had dermal filler injections within the last 12 months
12. Subjects who have had non-ablative laser treatments or IPL within the last 3 months
13. Subjects with known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs
14. Subjects currently using topically applied prescription medications on the face

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Change in Product tolerability | Change from Baseline at Day 42
  Product tolerability will be measured using the clinical grading of tolerance by evaluating the subjects reported local facial cutaneous tolerability including burning, stinging, and itching. Each scale will be measured with the following parameters, 0 = none (best possible outcome), 1 = mild, 2 = moderate, and 3 = severe (worst possible outcome). A decrease in scores or lack of significant increase indicates tolerability of the study treatment. The null hypothesis is that the mean change from baseline is zero.
Change in Product efficacy | Change from Baseline at Day 42
  Live Clinical Investigator grading of facial fine lines efficacy grading by using the modified Griffith's Photonumeric scale. The grading scale includes fine lines, crepiness, firmness, elasticity, smoothness, pore size, clarity, pigmentation, dark spot intensity, and skin tone evenness. The parameters for the scale are as follows, 0 = none (best possible outcome), 1 to 3 = mild, 4 to 6 = moderate, and 7 to 9 = severe (worst possible outcome). A decrease in scores indicates an improvement in study treatment efficacy. The null hypothesis is that the mean change from baseline is zero.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research
Locations (1):
- Austin Institute for Clinical Research, Inc., Pflugerville, Texas, United States